CLINICAL TRIAL: NCT01778244
Title: Metformin for Treatment of Antipsychotic-induced Dyslipidemia: a Randomized, Double-blind Study
Brief Title: Metformin for Treatment of Antipsychotic-induced Dyslipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Jingping Zhao, professor, Central South University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RRWu
Record Dates: First submitted 2013-01-19; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Dyslipidemia
Keywords: schizophrenia; dyslipidemia
MeSH Terms: conditions — Dyslipidemias; Schizophrenia | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin (Experimental): metformin
  Interventions: Drug: metformin
- placebo (Placebo Comparator): placebo

INTERVENTIONS:
Drug: metformin — 1000mg/day for 24 weeks
  Arms: metformin

SUMMARY:
Almost all antipsychotics can induce dyslipidemia, but no treatment has been established. Metformin can improve lipid levels in obese patients. The investigators conducted a randomized, placebo-controlled study to test the efficacy of metformin for antipsychotic-induced dyslipidemia.

DETAILED DESCRIPTION:
The study was designed as a double-blind randomized controlled trial, with research assessors and patients intended to be blind to the intervention status. The staff members performing the assessment were not involved in implementing any aspect of the intervention.162 patients were randomized to one of two 24-week individual treatments: metformin (1000mg/day)or placebo. Medications were provided in double-blind fashion.The assessments include lipid levels, body weight, body mass index, fasting glucose, fasting insulin and insulin resistance index.

ELIGIBILITY:
Inclusion Criteria:

Diagnostic and Statistical Manual of Mental Disorder-Fourth Edition (DSM-Ⅳ) criteria for schizophrenia dyslipidemia after antipsycotic treatment the duration of illness was less than 12 months taking only one antipsychotic stable outpatient the total score of Positive and Negative Syndrome Scale (PANSS)≤60.

-

Exclusion Criteria:

liver or renal diseases pregnant or lactating women cardiovascular diseases hypertension or diabetes mellitus

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
low-density lipoprotein cholesterol | 8 weeks

SECONDARY OUTCOMES:
high-density lipoprotein cholesterol | 8 weeks
adverse effects | 8 weeks

OTHER OUTCOMES:
body mass index | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Renrong Wu, MD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- Institute of Mental Health of The Second Xiangya Hospital, Central South University, Changsha, Hunan, China